CLINICAL TRIAL: NCT05717816
Title: Results of Hindfoot Fusion Using Modified Retrograde Intramedullary Femoral Nail With Plate in Diabetic Charcot Ankle Arthropathy : A Prospective Case Series Study
Brief Title: Hindfoot Fusion Using Intramedullary Nail in Diabetic Ankle Arthropathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ehab Ahmed Mohamed (Other)
Responsible Party: Sponsor-Investigator, Ehab Ahmed Mohamed, Participant investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: HFFIMN
Record Dates: First submitted 2022-12-22; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Charcot Arthropathy of Hindfoot
MeSH Terms: interventions — Fracture Fixation, Intramedullary; Bone Plates

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: intramedullary nail and plate — fusing Charcot ankle using retrograde intrameudllary femoral nail and plate

SUMMARY:
The aim of this study is to evaluate the outcome of healing rate of ankle fusion using modified retrograde IM femoral nail with plate in charcot ankle

DETAILED DESCRIPTION:
Charcot neuroarthropathy, is a progressive, noninfectious, and destructive joint disorder following trauma to a neuropathic extremity.The disorder mainly occurs in the foot and ankle joints. The process consists of bone and joint destruction, joint deformity, ulceration, and, if left untreated, may lead to amputation. The majority of the Charcot joint cases are associated with a neuropathic complication in patients with diabetes. Thus, with the increase in the current incidence of diabetes, the increase of Charcot joint cases is also expected.

The treatment of Charcot joint is variable including non operative, such as total contact casting, modified shoe, medication, and operative treatment. However, when the deformity is severe and unstable, the operative management is necessary. There are some surgical approaches to manage Charcot joint, such as exostectomy, Achilles tendon lengthening, arthrodesis with internal or external fixation, and amputation.

Arthrodesis is indicated in severe Charcot joint with significant instability. For Charcot ankle arthrodesis, internal fixation is more popular than external fixation in the absence of infection, significant bone defect, and poor soft tissue coverage. Some of the methods of internal fixation for ankle arthrodesis include the use of retrograde intramedullary nails, screws, and plates. many surgeons chose retrograde intramedullary nail fixation as the main method of internal fixation. However, limited compression and high nonunion rates have been found with intramedullary nail fixation.so using Plate with intramedullary nail will offer stiff constructs, more stability and better union rates. however, studies evaluating the use of combination fixation in the ankle arthrodesis for Charcot ankle, particularly nail with plate, are limited. [13] So, in this study the investigators will evaluate the outcomes of ankle arthrodesis using a combination of an intramedullary nail with plate in patients with diabetic Charcot ankle.

ELIGIBILITY:
Inclusion Criteria:

* Adult diabetic Patients who have (Brodsky type 2 and type 3A) Charcot ankle and HbA1c below 8

Exclusion Criteria:

* Prescence of active infection
* prescence of ulcers
* significant bone defect
* Vascular insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted at our trauma center at Assuit university hospital meeting the above mentioned criteria
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Radiological fusion | to be assessed up to one year post operative
  fusion of the Charcot ankle assessed by X- ray